CLINICAL TRIAL: NCT03370198
Title: An Open-label Dose Escalation Phase I Study to Assess the Safety and Clinical Activity of Multiple Hepatic Transarterial Administrations of NKR-2 in Patients With Unresectable Liver Metastases From Colorectal Cancer
Brief Title: Hepatic Transarterial Administrations of NKR-2 in Patients With Unresectable Liver Metastases From Colorectal Cancer
Acronym: LINK
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Difficulties in patient recruitment and clinical strategy modification based on new clinical data generated in the NKR-2 early development.
Sponsor: Celyad Oncology SA (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CYAD-N2T-004
Record Dates: First submitted 2017-11-08; First posted 2017-12-12 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Colon Cancer Liver Metastasis

STUDY DESIGN:
Intervention Model Description: There will be a hepatic transarterial administration of NKR-2 every 2 weeks for a total of 3 administrations within 4 weeks (28 days). Three dose-level will be assessed (dose escalation with 3 dose-levels or 3 cohorts).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dose-level 1 (Experimental): The dose-level 1 arm will use a 3+3 design. NKR-2 cells will be administered every 2 weeks (14 days) for a total of 3 administrations (hepatic transarterial administrations) within 4 weeks (28 days)
  Interventions: Biological: NKR-2 cells
- Dose-level 2 (Experimental): The dose-level 2 arm will use a 3+3 design. NKR-2 cells will be administered every 2 weeks (14 days) for a total of 3 administrations (hepatic transarterial administrations) within 4 weeks (28 days)
  Interventions: Biological: NKR-2 cells
- Dose-level 3 (Experimental): The dose-level 3 arm will use a 3+3 design. NKR-2 cells will be administered every 2 weeks (14 days) for a total of 3 administrations (hepatic transarterial administrations) within 4 weeks (28 days)
  Interventions: Biological: NKR-2 cells

INTERVENTIONS:
Biological: NKR-2 cells — NKR-2 cells will be administered (hepatic transarterial administration) every 2 weeks (14 days) for a total of 3 administrations within 4 weeks (28 days)
  Other Names: NKG2D CAR-T cells

SUMMARY:
The purpose of this study is to test an experimental anti-cancer immunotherapy called NKR-2 (modified T cells), to treat colorectal cancer with unresectable liver metastases. The trial will test three dose levels (dose escalation). At each dose, the patients will receive three successive hepatic transarterial administrations, two weeks apart, of NKR-2 cells. The study will enroll up to 18 patients.

ELIGIBILITY:
Inclusion Criteria:

* The patient must be ≥ 18 years old at the time of signing the ICF.
* The patient must have a histologically proven adenocarcinoma of the colon or rectum.
* The patient must have liver metastases non treatable with curative intent by surgical resection or local ablation at the time of registration.
* The patient must have measurable hepatic metastases defined by RECIST version 1.1 for solid tumors.
* The patient must have received one prior chemotherapy line for metastatic disease and have developed resistance or intolerance to this treatment.
* The patient must have an ECOG performance status 0 or 1.
* The patient must have the bone marrow reserve, hepatic and renal functions

Exclusion Criteria:

* Patients who are presenting evidence of ascites, cirrhosis, portal hypertension, main portal venous tumor involvement or thrombosis as determined by clinical or radiologic assessment.
* Patients who are planned to receive or concurrently receiving any non-cancer-directed investigational agent, or have received a non-cancer directed investigational agent within 3 weeks before the planned day for the first NKR-2 administration.
* Patients who are scheduled to receive concurrent growth factor (except erythropoietin), systemic steroid, other immunosuppressive therapy or cytotoxic agents (systemic or localized) other than the treatment authorized per protocol.
* Patients who underwent major surgery within 4 weeks before the planned day for the first NKR-2 administration.
* Patients who have received a live vaccine ≤ 6 weeks prior to the planned day for the first NKR-2 administration.
* Patients with a family history of congenital or hereditary immunodeficiency.
* Patients with history of any autoimmune disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2017-10-11 (Actual); Primary Completion 2018-01-15 (Actual); Study Completion 2018-12-15 (Actual)

PRIMARY OUTCOMES:
The occurrence of DLTs until 14 days after the last NKR-2 study treatment administration (Visit Day 43) | From study treatment start (Day 1) till 14 days after the last NKR-2 study treatment administration (Day 43)
  A DLT is defined as any Grade 3 or higher toxicity and any Grade 2 or higher autoimmune toxicity

SECONDARY OUTCOMES:
The occurrence of AEs and SAEs during the study treatment until 30 days after the last study treatment administration (Visit Day 57) | From study treatment start (Day 1) till 30 days after the last study treatment administration (Day 57)
  AEs and SAEs collection
The occurrence and duration of objective clinical response (complete response (CR), partial response (PR)) | through study completion (up to month 24)
  Complete response (CR), partial response (PR)
The occurrence and duration of clinical benefit (complete response (CR), partial response (PR) and stable disease (SD)) | through study completion (up to month 24)
  Complete response (CR), partial response (PR) and stable disease (SD)
The occurrence and duration of mixed response (MR) | through study completion (up to month 24)
  The different types of MR are defined according to the following criteria: at least 30% decrease in the longest diameter (or shortest diameter for nodal lesions) occurring in at least one target lesion recorded and measured at baseline. Such response occurring in otherwise SD or PD status of the sum of diameters of target lesions and without the appearance of one or more new lesions will be classified as "MR (SD)", which corresponds to a SD with target lesion regression or "MR (PD)", which corresponds to PD with target lesion regression and, the appearance of new lesion(s) in otherwise PR status of the sum of diameters of target lesions will be classified as "MR (PR)", which corresponds to a PR with new lesion.
The resection rate at Visits Day 57 and Month 3 | At visits Day 57 and Month 3
  Assessment of R0, R1 and R2 resections
The progression-free survival (PFS) | through study completion (up to month 24)
  The progression-free survival (PFS) is defined from registration in the study to the disease progression or death from any cause
The event-free survival (EFS) | through study completion (up to month 24)
  The event-free survival (EFS) is defined as the time from registration in the study to any of the following events: progression, local or distant recurrence, or death from any cause
The overall survival (OS). | through study completion (up to month 24)
  The overall survival (OS) is defined as the time from registration in the study to death. If death does not occur before the patient's last study visit, then the survival will be censored at the date when patient is known to be alive

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric Lehmann, MD, Principal Investigator — Celyad Oncology SA
Locations (1):
- Institut Jules Bordet, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No